CLINICAL TRIAL: NCT04077073
Title: Effects of Device-assisted Practice of Activities of Daily Living in a Close-to-normal Pattern on Upper Extremity Motor Recovery in Individuals With Moderate to Severe Stroke
Brief Title: Effects of Device-assisted Practice of ADL on Arm/Hand Recovery in Individuals With Moderate to Severe Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jun Yao, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00206913; R01HD095187 (NIH)
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: stroke rehabilitation; hand opening; flexion synergy; robot assisted treatment; functional electrical stimulation; motor recovery; brain plasticity
MeSH Terms: conditions — Stroke | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ReIn-hand and robot (Experimental): The participant will practice "reach, grasp, retrieve, and release (GR3)" a plastic jar for 40 trials per session, with the assistance of ReIn-hand to open their paretic hand and of robot to reduce the shoulder load.
  Interventions: Device: ReIn-Hand; Device: Robot
- ReIn-Hand (Active Comparator): The participant will practice "reach, grasp, retrieve, and release (GR3)" a plastic jar for 40 trials per session, with the assistance of ReIn-hand to open their paretic hand.
  Interventions: Device: ReIn-Hand

INTERVENTIONS:
Device: ReIn-Hand — ReIn-Hand assists the hand opening
  Other Names: ReIn-Hand assisted
Device: Robot — Robot supports the shoulder load
  Other Names: Robot support
  Arms: ReIn-hand and robot

SUMMARY:
A large number of post-stroke survivors cannot functionally use their paretic upper extremity (UE). This study therefore investigates effects of device-assisted practice of activities of daily living (ADL) in a close-to-normal pattern on UE motor recovery in individuals with moderate to severe stroke by measuring intervention-induced changes in clinical outcomes, UE kinematics, and functional and morphologic neuroplasticity. Positive findings may impact current clinical practice by pushing towards implementing device-assisted practice of ADLs and have the potential to benefit a large population.

DETAILED DESCRIPTION:
Thirty subjects for each group will be recruited. A REDCap database for this study will be setup to manage every step involved in the protocol. All the potential subjects will go through standardized steps:

1. Experienced research team members will conduct pre-screening of subjects from the Clinical Neuroscience Research Registry, which is maintained by the Physical Therapy and Human Movement Sciences (PTHMS) department at Northwestern University. Recruitment will also be conducted via flyers in various rehabilitation centers in the Chicagoland. The investigators will start the recruitment by an 'initial phone contact' to introduce the study and confirm the interests for participation. Once confirmed, a standardized 'phone screening' will be followed to partially go through the questions related to eligibility. Once passed all the questions over phone, a lab-based eligibility test will be scheduled at the department of PTHMS. During the first visit, the investigators will explain the study and answer all the related questions from potential participants. The paper consent form will be signed and dated by the individual once he/she agrees to participate, and a copy of the signed consent form will be given to the participant. Following consent, the blinded assessor will determine the eligibility using the inclusion and exclusion criteria.
2. The treating therapist will determine the settings of reliable and intuitive control of the paretic hand (ReIn-Hand) device. A 3D scan will be made to enable the produce of subject-specific ReIn-Hand device.
3. Qualified participants will undergo 2 baseline clinical assessments within 2 weeks.
4. All the enrolled participants will be randomly assigned to the either experimental or control group with the balance in Upper Extremity Fugl-Meyer Assessment (FMA) scores of the 2 groups. Randomization results will be concealed to the assessor all the time and will be only assessable to treating therapists and biostatisticians on the day for the first session of the assigned intervention.
5. The investigators will collect individual's magnetic resonance imaging (MRI) data and electroencephalogram (EEG) data within two weeks prior to the intervention. MRI scans will be performed at Northwestern University's Center for Translation Imaging. For EEG data collection, the investigators will first measure a subject's maximal voluntary torque (MVT) in the direction of shoulder abduction (SABD), maximum finger grasping forces of the paretic upper extremity (UE), maximum hand pentagon area, defined as the area formed by the tips of thumb and fingers, of the non-paretic hand when the hand is maximally stretched on a tabletop, and subject's upper- and forearm lengths for normalization purposes. For the hand opening task, participants' arm will be rested on the virtual table at the home position. Participants will relax in the home position for 5-7s and then to self-initiate maximal hand opening for 2s, without blinking or eye moving. For the hand opening with SABD loading, participants will perform the maximal hand opening while lifting the arm above table against 50% of his/her SABD MVT after 5-7s resting on the home position. A set of 60-70 trials will be collected for each condition, in a block randomized way (20-30 trials per block). Rest periods of ~15 s between trials and ~10 min between blocks will be included to avoid fatigue.
6. Intervention All participants will participate in a 24-session intervention, ~2 hours per session, 3 sessions per week, for 8 weeks in total. Research participants, training PTs, and clinical evaluators will be blind to group assignment.

   For all intervention, research participants will be seated with straps across the chest and waist to prevent unwanted trunk movement. The training technicians will stretch the paretic UE for up to 15 minutes. The ReIn-Hand device will be attached to the paretic UE and then positioned at a home position in 75° SABD, 30° shoulder flexion, and 60° elbow flexion.

   The first session will be a 'parameter adjusting session', during which the training PT will determine training parameters, including: 1) SABD load, 2) target(jar) distance, 3) jar width, 4) jar weight, 5) jar height, and 6) jar orientation. These training parameters will be established both on the table condition and using a robot. The robot modulates the supporting force in Z-direction applied to the arm while participants are required to lift the arm, thus changing the SABD load. The SABD load will be set as the maximum load that allows the participant to actively reach the target distance and achieve a ReIn-Hand mediated hand opening no less than 4 cm between the tips of the thumb and index fingers. After establishing SABD load, all the additional parameters (2-6) will be set, first with the established SABD load as following: Target distance is 70% of the distance of the max reach of the paretic UE when fully supported on a frictionless table created by the robot; Jar width will be increased in 0.5 cm increments, by adding padding around the jar, to the max width the participant can achieve with the ReIn-Hand; Jar height (i.e., distance from the lowest part of the jar to the surface of the table) will be set as 2 cm increments to the max height the participant can successfully (and painlessly) reach the jar; Jar orientation (i.e., the relation of the long axis of the jar to the table surface) will be set as 2° increments to the maximum amount that allows the participant to successfully grasp the jar; and Jar weight will be increased in 100 g increments, stopping if the participant experiences pain or cannot lift the jar. The Training PT will then repeat the steps 2-6 to determine these parameters (2-6); however, this time without robot support and thus using a height-adjustable table.

   Once the intervention parameters are set, the training technician will guide the participant to perform 'reaching-grasping-retrieving-and- releasing' (GR3) activities using these parameters. Participants in the experimental group will be trained using the robot. Their forearm of a participant will be attached to an orthosis, which will be firmly attached to the robot. Participants in the experimental group will be trained on a regular table. All training sessions will consist of 40 trials (about 1 hour) of GR3 activities, which include: 1) Reaching towards a plastic jar (diameter=3cm, weight=30g when empty); 2) Activating finger/wrist extensor muscles to trigger the ReIn-Hand device, which in turn assists the opening of the paretic hand while reaching; 3) Grasping the jar; 4) Retrieving the jar to the home position and placing it on the table; and 5) Releasing the jar. To avoid fatigue, a resting time of 20-30 seconds will be provided between trials. Participants in the control group will be encouraged to perform GR3 activities with the arm above the table.

   A successful trial requires the completion of all five tasks required during one trial: Reaching towards a plastic jar, triggering the ReIn-Hand device, grasping the jar, retrieving the jar to the home position, and placing it on the table, and releasing the jar. An unsuccessful trial is defined as the failure to complete one of the five tasks during one trial. The result of each of the 40 trials will be recorded by the training technician.

   The Training PT will review the training performance after each session to determine if adjustment of parameters is necessary for the next session. If a participant successfully completes 30/40 trials in 2 successive sessions, the training PT will re-adjust all the parameters at the following session to progressively challenge the participant. New parameters then will be implemented by the training technician during the following session.
7. Weekly outcome measures. The blinded clinical assessor will measure the following outcomes weekly: Box and Blocks Test, Quantitative Measure of Hand Opening and Closing, and Cutaneous Sensory Touch Threshold.
8. The blinded clinical assessor will check participant's sensory and motor function using the same clinical assessments as that used for baseline within 1 week after the intervention.
9. Within one week after the end of intervention, the investigators will repeat the neural imaging and biomechanical data collection, using the same protocols as stated before.
10. Three-month follow-up. Three months after the intervention, the blinded clinical assessor will check participant's sensory and motor function using the same clinical assessments as stated before. To maximize the retention, the investigators will have a clear and standardized communication of our expectations of the participant over the course of the study. For each participant, the project coordinator will generate a personal timetable with scheduling of experiments. Flexibility of appointments will be included. Finally, the project coordinator will call the participants about at 7 days and then 1 day before the scheduled 3-month follow up to remind the last assessment.

AE and SAE reporting Adverse event (AE) report form has been implemented in the RedCap database, which can be used at any time. The investigators will report all AEs to the Northwestern Institutional Review Board (IRB) per established policies and requirements. The investigators will create AE reports every six months to review for trends and troubleshoot any issues that arise and require study protocol revision. If any AEs are reported that require follow-up medical care, the investigators will immediately refer the participant back to his/her physician team.

Serious adverse events (SAEs) that are unanticipated, serious, and possibility related to the study intervention will be reported to the Independent Monitor(s), IRB, and National Institute of Child Health and Human Development (NICHD) in accordance with requirements. Unexpected fatal or life-threatening AEs related to the intervention will be reported to the Northwestern IRB in accordance with IRB requirements within 24 hours, and to the NICHD program Officer with 7 days. Other serious and unexpected AEs related to the intervention will also be reported to the Northwestern IRB in accordance with IRB requirements within 24 hours, and to the NICHD program Official within 15 days. Anticipated or unrelated SAEs will be handled in a less urgent manner but will be reported to the Independent Monitor(s), IRB, NICHD, and other oversight organizations in accordance with their requirements. In the annual AE summary, the Independent Monitor(s) Report will state that they have reviewed all AE reports.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21-80
2. Paresis confined to one side, with substantial motor impairment of the upper limb and some residual voluntary movement (UE FMA in the range of 10-40/66, CMSA_H stage of the hand section <=4)
3. Capacity to provide informed consent
4. Ability to elevate their limb against gravity up to at least 75 degrees of shoulder flexion and to generate some active elbow extension
5. Ability to open hand with a thumb-to-index finger distance ≥4 cm, with the assistance of the ReIn-Hand device with the help of a physical therapist
6. MRI compatible
7. Discharged from all forms of physical rehabilitation
8. Intact skin on the hemiparetic arm
9. Be tolerate sitting for no less than 1 hour
10. Montreal Cognitive Assessment (MoCA) score >=23

Exclusion Criteria:

1. Motor or sensory impairment in the non-affected limb
2. Any brainstem and/or cerebellar lesion
3. Severe concurrent medical problems (e.g. cardiorespiratory impairment, uncontrolled hypertension, inflammatory joint disease)
4. History of neurologic disorder other than stroke (Parkinson's Disease, Acute Lateral Sclerosis, Multiple Sclerosis, Traumatic Brain Injury, peripheral neuropathy, Amyotrophic lateral sclerosis, spinal cord injury, Dementia)
5. Any acute or chronic painful condition in the upper extremities or spine, indicated by a score ≥5 on a 10-point visual analog scale
6. Using cardiac pacemaker, implanted cardioverter defibrillator, neurostimulation system inside the brain or spinal cord, bone growth box fusion stimulation
7. Seizure in the last 6 months
8. Severe upper extremity sensory impairment indicated by absent sensation on the tactile sensation subscale (light touch and pressure items) of the Revised Nottingham Assessment of Somato-Sensations (score<4)
9. Chemo denervation: botulinum toxin, dysport, or Myobloc or phenol block injection to any portion of the paretic UE within the last 6 months, or phenol/alcohol injections <12 months before participation
10. Unable to passively attain 90 degrees of shoulder flexion and abduction, measured using a goniometer based on adapted methods
11. Flexion contractures larger than 45 degrees in the elbow, wrist, metacarpophalangeal joints (MCP) and interphalangeal joints (IP) of thumb and index finger
12. Pregnant or planning to become pregnant
13. Participating in any experimental rehabilitation or drug studies
14. Inability to attend intervention sessions 3 times a week during 8 weeks, as well as to assessments/evaluations and follow up
15. Upper extremity musculoskeletal impairment limiting function prior to stroke
16. Currently using oxygen
17. Upper limb amputation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Box and Blocks Test (BBT) from baseline to 1 week post-intervention | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time per week during intervention, 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up
  Individuals are seated at a table, facing a rectangular box that is divided into two square compartments of equal dimensions by means of a partition. One hundred and fifty small wooden cubes or blocks are placed in one compartment or the other. The individual is instructed to move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds. The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period. Patients hand must cross over the partition in order for a point to be given, and blocks that drop or bounce out of the second compartment onto the floor are still rewarded with a point. Multiple blocks carried over at the same time count as a single point.

SECONDARY OUTCOMES:
Change in Quantitative measure of hand opening area and closing force | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time per week during intervention, 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up
  Individual will be instructed to rest paretic hand on a cylinder that is covered with an array of pressure sensors (Pressure Profile Systems, Inc., Los Angeles, CA 90045). Furthermore, 5 markers (9x9 mm) with unique optical features will be placed on the tip of the thumb and the 4 fingers. Individual will then be instructed to perform following task in their comfortable pace: 1) resting, 2) maximally open the paretic hand, and 3) maximally close the paretic hand against the cylinder. Position (with an accuracy of 1mm) and angular (with an accuracy at 0.02 degree) information of fingertips will be captured by 2 registered portable Moire Phase Tracking cameras (Metria Innovation, Inc., Wauwatosa, WI); and the flexion force under the 4 fingers and thumb will be measured by the pressure sensors. This will allow for tracking of the hand pentagon area and closing force during intervention.
Change in Cutaneous Sensory Touch Threshold using Semmes-Weinstein Monofilaments | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time per week during intervention, 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up
  The monofilament test is a threshold assay used to determine the minimum stimulation that can be felt by a subject.
Change in Upper extremity Fugl-Meyer Assessment Score | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up.
  The Fugl-Meyer Assessment of Motor Recovery after stroke evaluates and measures motor impairment in post-stroke hemiplegic patients. Different movements are judged on the individuals ability to perform with full capacity, limited capacity, or total inability to complete the required movements. We will use the upper extremity part of FMA, with scores ranging from 0-66, 0 and 66 representing no and normal residual upper extremity motor function, respectively.
Change in Sensory Assessment (Stereognosis) | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up
  The individual will be asked to use their paretic hand to identify a number of everyday items through touch alone. Scores range from 0-24, with 24 indicating full stereognosis function and 0 representing complete absence of stereognosis.
Change in Stroke Impact Scale (SIS) | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up.
  The SIS is a 59 item measure of strength, hand function, activities of daily living, mobility, communication, emotion, memory, and participation. Each item is rated in a 5 point scale in terms of difficulty experienced in completing the item, ranging from 1 (could not do it at all) to 5 (not difficult at all)
Change in Motor Activity Log (MAL) | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up.
  It is a semi-structured interview to assess arm function. Individuals are asked to rate quality of movement and amount of movement during 30 daily functional tasks., including object manipulation as well as the use of the arm during gross motor activities. Items scored on a 6-point ordinal scale, with 0 representing never and 6 as normal.
Change in Action Research Arm Test (ARAT) | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up.
  The ARAT test is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). ARAT is a validated quick assessment of the paretic arm's functional disabilities, which offers uncomplicated and comprehensive feedback on the function of their arm, hand and fingers. Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points indicating better performance.
Change in Chedoke McMaster Stroke Assessment (CMSA) Hand Subscale | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up.
  This test evaluates the stage of motor recovery for the paretic hand. Scores range from 0-7, with 7 representing full function of the hand.
Change in Revised Nottingham Sensory Assessment: Kinaesthesia Subscale | This will be measured twice pre-intervention (within 1 week prior to intervention), 1 time immediately after conclusion of intervention (within 1 week), and 1 time at the 3 month follow up.
  The kinaesthesia subscale measures an individual's ability to sense movement, direction of movement, and position sense at a given joint. The assessment involves the tester initiating passive movement in the individuals affected finger, wrist, elbow, and shoulder; while the individual attempts to match those movement with their opposite extremity. Scores for each joint range from 0-3, with 3 representing intact position, direction, and sense of movement.
Change in Coupling forces generated by shoulder and elbow while opening hand with or without lifting | This will be measured 1 time pre-intervention (within 1 week prior to intervention), and 1 time immediately after conclusion of intervention (within 1 week).
  This metric quantifies the coupling forces (during hand opening without lifting) or movements (during hand opening and lifting) generated by shoulder and elbow.
Change in Hand pentagon area (HPA) while opening with or without lifting | This will be measured 1 time pre-intervention (within 1 week prior to intervention), and 1 time immediately after conclusion of intervention (within 1 week).
  This metric quantifies the areas formed by the thumb and fingertips during maximally opening the paretic hand with or without lifting.
Change in Laterality Index for the cortical activity related to hand opening | This will be measured 1 time pre-intervention (within 1 week prior to intervention), and 1 time immediately after conclusion of intervention (within 1 week).
  Laterality Index is defined as (LI = (I-C)/(I+C)), where 'I' and 'C' are the current density strengths from the ipsilesional and contralesional sensorimotor cortices (i.e., combined primary sensorimotor and secondary motor cortices). LI reflects the relative contributions of each cerebral hemisphere to the source activity, with a value close to +1 for an ipsilesional source distribution and -1 for a contralesional source distribution.
Change in Cortical activity ratio (CAR) | This will be measured 1 time pre-intervention (within 1 week prior to intervention), and 1 time immediately after conclusion of intervention (within 1 week).
  The cortical activity ratio is defined as the ratio between the sum of the current density strength of nodes in one of the regions of interest (ROI), to the sum of current density strength of nodes in the whole sensorimotor cortices. The CAR reflects the relative strength from one ROI as normalized by the total combined strength of the 4 ROIs.
Change in Gray matter (GM) density | This will be measured 1 time pre-intervention (within 1 week prior to intervention), and 1 time immediately after conclusion of intervention (within 1 week).
  It quantifies the gray matter density, which in a particular region of the brain appears to correlate positively with various abilities and skills.
Change in Fractional anisotropy (FA) of bilateral cortico-fugal tracks | This will be measured 1 time pre-intervention (within 1 week prior to intervention), and 1 time immediately after conclusion of intervention (within 1 week).
  It quantifies the white matter integrity of the targeted motor descending tracks.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yao, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - 645 N Michigan Ave, Suite 1100, Chicago, Illinois
  - Northwestern University, Dept. of PTHMS, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drogos JM, Carmona C, Arceo R, Yao J. Effects of device-assisted practice of activities of daily living in a close-to-normal pattern on upper extremity motor recovery in individuals with moderate to severe stroke: study protocol of a randomized control trial. Trials. 2025 Jul 4;26(1):238. doi: 10.1186/s13063-025-08930-7. PMID 40616111
- [Derived] Carmona C, Sullivan JE, Arceo R, Drogos J, Besser S, Gutierrez S, Jeteric Z, Wyman J, Yao J. Development and Preliminary Validity Study of a Modified Version of the Upper Extremity Fugl-Meyer Assessment for Use in Telerehabilitation. J Neurol Phys Ther. 2023 Oct 1;47(4):208-216. doi: 10.1097/NPT.0000000000000447. Epub 2023 Jun 14. PMID 37314323

DOCUMENTS (2):
  • Study Protocol (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT04077073/Prot_006.pdf
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT04077073/ICF_007.pdf